CLINICAL TRIAL: NCT00362804
Title: Augmentation of Antipsychotic Partial Responders With Tetrabenazine
Brief Title: Tetrabenazine for Partial Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Gary Remington, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 240/2001
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: tetrabenazine; partial response; psychosis; schizophrenia; schizoaffective disorder; partial response to antipsychotics
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Tetrabenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tetrabenazine — The initial TBZ dose will be 12.5 mg and the dose will be increased to 25 mg at Week 2. Thereafter, the dose can be decreased to 12.5 mg or increased in 12.5 mg increments at weekly intervals, depending on clinical response and tolerability, to a maximum of 75 mg/day. For 37.5 and 50 mg daily, administration will be BID i.e., 25 mg QAM, 12.5 or 25 mg QHS. For 62.5 or 75 mg daily, a TID dosing will be employed i.e., 25 mg QAM, 12.5 or 25 mg QPM, 25 mg QHS

SUMMARY:
Purpose of Study:

A) To improve outcome in large population of antipsychotic patients with schizophrenia or schizoaffective who are only partial responders B) To increase understanding of pharmacology and mechanisms of action underlying antipsychotic effect

Hypothesis/Objectives of the Study:

Tetrabenazine, through its pre-synaptic action, should augment the post-synaptic effects of an antipsychotic.

Background and Rationale for the study:

Preliminary evidence that other amine-depleting agents e.g., reserpine, can induce such an effect

DETAILED DESCRIPTION:
Since the 1950's, antipsychotics have been used as the mainstay treatment to control symptoms of schizophrenia. However, soon after their introduction it became apparent that a substantial number of individuals show a less than optimal response to these drugs - as many as 30% of schizophrenics using conventional antipsychotics derive little benefit. Furthermore, 'atypical' generation antipsychotics such as clozapine which proves to be the most beneficial for partial responders and represents the cornerstone of treatment-resistant schizophrenia, offers a response rate as low as 30% in those showing an inadequate response. Moreover, many individuals decline clozapine as an option, or cannot tolerate it.

For these reasons, augmentation strategies play an important role in the treatment of antipsychotic partial responders. We have systematically reviewed the different augmentation options, and reached the conclusion that most such strategies are theoretically speculative and empirically unsupported.

At the same time though, we recognize that augmentation strategies are common practice in the clinical setting. With so many individuals showing only a partial response to antipsychotic treatment (typical or atypical), it has become a practical reality in efforts to offer further improvement. Often, this come in the form of adding one or even more antipsychotics, although the evidence for such an approach is less than compelling and neuroimaging from our centre has cautioned against this approach.

With a variety of other potential augmentation strategies available, we have chosen to focus on tetrabenazine (TBZ), which is currently licensed here in Canada for the management of hyperkinetic movement disorders.

The choice of TBZ as an augmentation strategy arises from several lines of investigation:

* TBZ, like reserpine, is a pre-synaptic monoamine-depleting agent or inhibitor of vesicular monoamine transporter, and hence will act to dampen abnormal dopamine release in patients already on a primary post-synaptic D2 blocking compound, as is the case (to varying degrees) with all antipsychotics currently available.
* There are anecdotal reports with reserpine, indicating that it can augment response in patients showing only a partial response to antipsychotic (atypical, as well as typical) partial responders.
* TBZ appears to have a low-affinity post-synaptic D2 effect, still well below the 80% threshold where one begins to see motor side effects.
* TBZ has inherent anti-dyskinetic properties, thereby offering an additional secondary benefit.

We are proposing to carry out a controlled double-blind trial, using TBZ off-label in patients with schizophrenia or schizoaffective disorder only partially responsive to antipsychotics. We feel that the choice of this approach is empirically sound and, in fact, offers advantages to the more common approach of adding several antipsychotics. Our decision to maintain out focus on the dopaminergic system arises from the growing body of evidence that dopamine blockade, particularly at the level of the D2 receptor, is central to antipsychotic activity, in combination with the lack of current evidence supporting the distinct advantages of incorporating other systems.

Given the limited success with augmentation strategies in schizophrenic patients to date, any evidence of efficacy and safety with this combination will add considerably to options that might be considered in the clinical setting. This same information could also prove very useful in shaping investigations related to the pharmacology of schizophrenia and development of future compounds.

ELIGIBILITY:
Inclusion Criteria:

* has been on an antipsychotic medication for at least 3 months and achieved the maximum dose vis à vis tolerability/side effects.
* Partial response to antipsychotic medication (CGI > 4; BPRS [Anchored, 18-item] total > 30; single item score > 4 on 2 positive symptom items)
* has been on at least 2 previous antipsychotic trials of 4-6 weeks in duration at a dose reaching 400-600 mg chlorpromazine (or equivalent) with no clinical improvement

Exclusion Criteria:

* age < 18 or > 65
* previous documentation of hypersensitivity to tetrabenazine
* SCID criteria for a current depressive episode
* MAOI administration within 2 weeks of tetrabenazine treatment
* concomitant desipramine use
* diagnosis of idiopathic Parkinson's disease and/or levodopa treatment
* current unstable medical illness and current substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-02; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
BPRS | weekly assessments
CGI | weekly assessment

SECONDARY OUTCOMES:
GAF/NOISE | weekly
SAS | weekly
AIMS | weekly
BAS | weeekly
UKU (a general measure of adverse effects) | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Gary Remington, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada